CLINICAL TRIAL: NCT01316536
Title: Music Therapy is Associated With Decreased Pain and Agitation in Intubated ICU Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inability to recruit participants despite numerous attempts
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: H9025-35126-01; 10-04501 (Other: UCSF CHR)
Record Dates: First submitted 2011-03-14; First posted 2011-03-16 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Music Therapy for Pain and Sedation
Keywords: pain, agitation, music
MeSH Terms: conditions — Pain; Psychomotor Agitation | interventions — Sound

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- With Music (Experimental): This randomized group will receive music
  Interventions: Other: provide headphones with music playing
- Control Arm (Placebo Comparator): Will not receive music but will receive audio loop of recorded ICU sounds
  Interventions: Other: Sounds

INTERVENTIONS:
Other: provide headphones with music playing — Participants will be provided with music through headphones
  Arms: With Music
Other: Sounds — recorded ICU sounds will be provided to participants through headphones
  Arms: Control Arm

SUMMARY:
The study is designed to analyze the use of music therapy to decrease pain and agitation in intubated ICU patients.

DETAILED DESCRIPTION:
This is a randomized, prospective single-blinded placebo-controlled study of consecutive intubated ICU patients requiring anxiolytics and analgesic medications. Patients will be randomized into two groups: one group will receive music (MUSIC), whereas the other group (CONTROL) will wear headphones, but hear an audio loop of recorded ICU sounds (vent alarms, ambient noise, talking, etc). The two groups will then be analyzed for sedation and analgesia requirements; Ramsay sedation score, ICP in brain injured patients, ventilator days, ICU length of stay, hospital length of stay, mean arterial blood pressure (MAP).

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 70 years old, requiring intubation andmechanical ventilation, requiring sedation with propofol or benzodiazepines and/or analgesia with narcotics

Exclusion Criteria:

* hearing loss, psychiatric illness, hemodynamically unstable (requirement for vasopressor support)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Decreased sedation and pain requirements | maximum of 7 days from study entry while still intubated and sedated

SECONDARY OUTCOMES:
ICU length of stay | from admission date to ICU to discharge date from ICU while on study

CONTACTS AND LOCATIONS:
Overall Officials: Julin Tang, MD, Principal Investigator — University of California, San Francisco; Dante Yeh, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco at San Francisco General Hospital, San Francisco, California, United States